CLINICAL TRIAL: NCT02763891
Title: Effect of Body Suspension and Tilting Exercises in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 555
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson Disease
Keywords: Balance; Mobility; Trunk control
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Subjects submitted to a 30-minute session of suspension and tilting exercises on the Chordata equipment (PI: 0804871-1 and BR 10 2012 009901-2) twice a week for eight weeks.
  Interventions: Other: Intervention group (Body body suspension and tilting exercises)
- Control group (Sham Comparator): Subjects submitted to a 30-minute passive muscle stretching session twice a week for eight weeks.
  Interventions: Other: Control group (global muscle stretching)

INTERVENTIONS:
Other: Intervention group (Body body suspension and tilting exercises) — The body suspension and tilting exercise program (Chordata Method) involved suspending the body in the apparatus while performing tilting exercises. The Chordata apparatus consists of a steel structure with special springs and a harness specifically manufactured for practicing the Chordata Method. During the training sessions, the prescribed exercises emphasize the repetition of movements designed to promote different types of muscle contractions (concentric, eccentric, static) performed in different body positions and joint angles. Thus, when using the method, patients experience maximal functional performance beyond to the body mass centre, activating trunk antagonist muscles and motor memory evocation. Each session lasts 30 minutes.
  Other Names: Chordata body suspension and tilting
  Arms: Intervention group
Other: Control group (global muscle stretching) — Subjects receiving submitted a global muscle stretching session twice a week for eight weeks. During this period. All participants are requested to don't engage in any additional type of exercise program or physical activity throughout the study period.
  Other Names: Control
  Arms: Control group

SUMMARY:
This study evaluates the effect of body suspension and tilting exercises (performed in Chordata apparatus) on the balance and mobility of subjects with Parkinson disease. Half of patients will perform the exercise protocol while the other half will receive passive muscle stretching and maintain the usual routine.

DETAILED DESCRIPTION:
Body suspension and tilting exercises performed in the Chordata equipment might be an effective option to improve trunk muscles activation and to facilitate functional balance and mobility control in Parkinson's disease (PD). To evaluate this hypothesis, subjects will be randomized into control group or intervention group. Intervention group will receive 30-minute session of body suspension and tilting exercises on the Chordata equipment (PI: 0804871-1 and BR 10 2012 009901-2) twice a week for eight weeks, while the control group will receive passive muscle stretching and maintained their usual routine during the same period. Both groups will be assessed at baseline and immediately after the intervention protocol. Finally, a follow-up evaluation will be performed 8 weeks after the protocol ending (to verify possible long-lasting effects of this exercise protocol).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to go to training or assessment places;
* Subjects that are agreement with the study protocol and sign the ;
* Subjects in stage I, II or III of Parkinson disease according to the Hoehn and Yahr scale.

Exclusion Criteria:

* Subjects do not keep their usual routine (apart of the research protocol);
* Subjects with physical or functional limitations that prevent the assessment test battery;
* Subjects with heart or lung diseases that prevent the exercise performance;
* Subjects with cancer;
* Subjects with major visual deficits;
* Subjects with recurrent vertigo;
* Subjects with uncontrolled systemic blood pressure.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | At 8th week (in the end of exercise protocol).
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The person wears regular footwear and customary walking aid.

SECONDARY OUTCOMES:
Berg Balance Test | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  The Berg Balance Scale (BBS) is a widely used clinical test of a person's static and dynamic balance abilities. For functional balance tests, the BBS is generally considered to be the gold standard. The test takes 15-20 minutes and comprises a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.
Functional Reach Test | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  The Functional Reach test can be administered while the patient is standing. The patient is instructed to next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the 3rd metacarpal head on the yardstick. Instruct the patient to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is recorded in centimetre (cm). Scores are determined by assessing the difference between the start and end position is the reach distance. Three trials are done and the average of the last two is noted.
Baropodometry (Stabilometric parameters) | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  In the test protocol adopted data uptake of the examination will be assessed walking on the pressure platform (dynamic measure) and stopped on the pressure platform with opened eyes (static measure).
Unified Parkinson Disease Rating Scale (UPDRS) | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  The UPDRS is a rating tool to follow the longitudinal course of Parkinson's Disease. It is made up of the 1) Mentation, Behavior, and Mood, 2) ADL and 3) Motor sections. These are evaluated by interview. Some sections require multiple grades assigned to each extremity. A total of 199 points are possible. 199 represents the worst (total) disability), 0--no disability.
Parkinson's Disease Questionnaire (PDQ-39) | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  The Parkinson's Disease Questionnaire (PDQ-39) is primarily used in clinical trials of therapeutics intended to benefit individuals with Parkinson's disease.
Timed Up and Go Test | At baseline, at 8th week (in the end of exercise protocol) and at 16th week (follow-up).
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The person wears regular footwear and customary walking aid. The investigators will measure the "change" at different time frames.

OTHER OUTCOMES:
Hoehn and Yahr Staging of Parkinson's Disease | This test will be performed just at baseline (to classify the subjects).
  The Hoehn and Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress.

CONTACTS AND LOCATIONS:
Overall Officials: Irênio G da Silva Filho, PhD, Study Chair — Pontifícia Universidade Católica do Rio Grande do Sul; Carlos Roberto M Rieder, PhD, Study Chair — Hospital de Clínicas de Porto Alegre; Régis G Mestriner, PhD, Study Director — Pontifícia Universidade Católica do Rio Grande do Sul; Charlene B de Oliveira, MSc, Principal Investigator — Pontifícia Universidade Católica do Rio Grande do Sul
Locations (1):
- Serviço de Neurologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided